CLINICAL TRIAL: NCT02068092
Title: A Pilot Study of Hydroxytyrosol, a Component of Olive Oil for Breast Cancer Prevention In Women At High Risk Of Breast Cancer
Brief Title: Olive Oil for High Risk Breast Cancer Prevention in Women
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Jenny C. Chang, MD, Principal Investigator, The Methodist Hospital Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00009472; 0713-0108 (Other: HMRI IRB)
Record Dates: First submitted 2014-02-18; First posted 2014-02-21 (Estimated); Results first posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — 3,4-dihydroxyphenylethanol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Hydroxytyrosol (Experimental): Hydroxytyrosol 25 mg orally once daily for 1 year.
  Interventions: Drug: Hydroxytyrosol

INTERVENTIONS:
Drug: Hydroxytyrosol

SUMMARY:
This is a pilot study evaluating the effect of hydroxytyrosol, a component of olive oil, on mammographic density in women at high risk of developing breast cancer.

DETAILED DESCRIPTION:
This is a pilot study evaluating the effect of hydroxytyrosol, a component of olive oil, on mammographic density in women at high risk of developing breast cancer. Participants will take hydroxytyrosol orally once daily for 1 year. Breast density as determined by mammography and the safety/toxicity of hydroxytyrosol will be assessed.

ELIGIBILITY:
Inclusion Criteria

1. Female aged ≥18 years of age.
2. Elevated risk of breast cancer as defined by at least one of the following categories and have declined tamoxifen and/or raloxifene therapy:

   1. Diagnosis of lobular carcinoma in situ (LCIS), atypical ductal, or lobular hyperplasia.
   2. A known deleterious mutation in BRCA1, BRCA2, PTEN, or TP53. (Note: The participant must be a documented carrier to meet this criterion. If there is a known mutation in a hereditary breast cancer susceptibility gene in a participant's family member, the participant herself must have undergone genetic testing as per National Comprehensive Cancer Network guidelines to be eligible per this criterion.)
   3. Modified Gail/CARE model risk at 5 years ≥ 1.67%. (Note: Risk models are to be used only if there is no known previous diagnosis of resected ductal carcinoma in situ [DCIS] or LCIS and there is no known deleterious mutation in BRCA1, BRCA2, PTEN, or TP53)
   4. 10% or more probability of BRCA mutation by BRCAPRO or similar model
3. Must have at least one breast available for imaging and biopsy. A previously irradiated breast (i.e., for resected DCIS) is not evaluable for breast imaging or biopsy.

   a. Allow for submission of core needle breast material for future use.
4. Baseline mammogram performed within 90 days prior to study entry, done on a digital mammography machine, that are reported as normal or benign.
5. Baseline mammographic density > 10% based upon the classification system (2 = 11-50%, "scattered fibroglandular densities"; 3 = 51-75%, heterogeneously dense; 4 = >75%, extremely dense). Women with a baseline mammographic density of ≤ 10% (1 = ≤10%, breasts are almost entirely fat) will not be eligible
6. Eastern Cooperative Oncology Group performance status of 0-1.
7. Prior anticoagulant therapy use is allowed provided therapy is discontinued at least 7 days prior to the breast biopsy in order to reduce the risk of bleeding. For participants who have taken an anticoagulation within the past 7 days, international normalized ratio must be ≤ 1.5 x institutional upper limit of normal and prothrombin time and partial thromboplastin time ≤ ULN prior to the breast biopsy.
8. Must agree to use effective consistent contraception. Hormone-based birth control (pills, patches, or shots) is allowed. Hormone replacement therapy is not allowed for postmenopausal participants.
9. Must not participate in any other clinical trial for the treatment or prevention of cancer unless they are no longer receiving the intervention and are in the follow-up phase only. Participants must also agree not to join such a trial while participating in this study.
10. Provide written informed consent.

Exclusion Criteria

1. DCIS or previous invasive ductal carcinoma.
2. Any prior malignancy except for the following: adequately treated basal cell or squamous cell skin cancer and in situ cervical cancer.
3. Prior tamoxifen or raloxifene use in the past 1 year.
4. Pregnant or breastfeeding.
5. Bilateral breast implants. Prior breast reduction surgery is allowed.
6. Mammograms that are reported as suspicious.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Chang, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (3):
- United States (3):
  - Houston Methodist Hospital, Houston, Texas
  - Houston Methodist Hospital Willowbrook, Houston, Texas
  - Houston Methodist Hospital Sugar Land, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No
To be determined

REFERENCES:
- [Derived] Puri A, Yin Z, Granados-Principal S, Ensor J, Guzman L, Rosato R, Zhao H, Wong S, Wang L, Patel T, Chang JC. Hydroxytyrosol, a Component of Olive Oil for Breast Cancer Prevention in Women at High Risk of Cancer. Int J Breast Cancer. 2025 Jan 21;2025:8831168. doi: 10.1155/ijbc/8831168. eCollection 2025. PMID 39882028

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Hydroxytyrosol
Started | 51
Completed | 41
Not Completed | 10
Not completed — Physician Decision | 2
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 4
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Groups:
- Hydroxytyrosol: Hydroxytyrosol 25 mg orally once daily for 1 year.
  Hydroxytyrosol
Arm/Group | Hydroxytyrosol
Number analyzed (Participants) | 51
Age, Customized [Median (Full Range); unit: years]
  Median Age | 54 [35 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Caucasian | 41
  African American | 4
  Asian | 2
Menopausal Status [Count of Participants; unit: Participants]
  Pre-menopausal | 22
  Post-menopausal | 29

OUTCOME MEASURES:

1. Primary Outcome: Change in Maximum Volumetric Breast Density Percentage
Description: Change in Maximum Volumetric Breast Density Percentage from Baseline at 12 Months. Maximum volumetric breast density (max VBD%) which is calculated by fibroglandular breast volume divided by total breast volume (checked on the higher side, left or right) was used to obtain the study's endpoints. The primary endpoint was the annualized percent decrease in max VBD% between baseline (BL) and end-of-treatment (EOT) with HT.
Time Frame: Baseline and 12 months
Population: There were 26 patients who had both baseline and end of treatment raw images of mammograms available on which quantitative analysis using volpara software was performed.
Measure: Mean (95% Confidence Interval); unit: Mean decrease in max VBD percentage
Arm/Group | Hydroxytyrosol
Number analyzed (Participants) | 26
Mean decrease in max VBD percentage | -0.038 [-0.112 to 0.035]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with adverse events as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events v4.03
Time Frame: From informed consent up to 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Hydroxytyrosol
Number analyzed (Participants) | 51
Participants | 2

3. Other Pre Specified Outcome: Expression of Ki67 in Tumor Tissue
Description: To determine the expression of Ki67 in tumor tissue
Time Frame: From baseline and at 12 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: MRI Breast Density
Description: To determine breast density as assessed by magnetic resonance imaging
Time Frame: From baseline and at 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse events that begin or worsen after informed consent will be continuously recorded on months 3, 6, and 12 and 13 (Days 90, 180, 360 and 390 (+/- 14 days for each assessment) up until at least 30 days after the last dose of study treatment.
Arm/Group | Hydroxytyrosol
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 2/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hydroxytyrosol (N=51)
Fatigue (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/92/NCT02068092/Prot_SAP_000.pdf